CLINICAL TRIAL: NCT05867121
Title: A Phase Ib, Open-label, Multicenter Dose-expansion Study Evaluating the Safety, Pharmacokinetics, and Activity of RO7496353 in Combination With a Checkpoint Inhibitor With or Without Standard-of-care Chemotherapy in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, & Activity of RO7496353 in Combination With a Checkpoint Inhibitor With or Without Standard-of-care Chemotherapy in Participants With Locally Advanced or Metastatic Solid Tumors; Urothelial Carcinoma Substudy in Association With RO7496353 Study GO44010
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO44010; 2022-502615-11-00 (EU CTIS Number)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer; Gastric Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Carcinoma, Transitional Cell | interventions — atezolizumab; Capecitabine; S 1 (combination); Tegafur; Nivolumab; Oxaliplatin; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: NSCLC (Experimental): Participants with NSCLC will receive RO7496353, and atezolizumab, given as an intravenous (IV) infusion at an assigned dose on Day 1 of each 21-day cycle until unacceptable toxicity or symptomatic deterioration attributed to disease progression (PD).
  Interventions: Drug: RO7496353; Drug: Atezolizumab
- Cohort B: GC (Experimental): Participants with GC will receive RO7496353, nivolumab, and oxaliplatin, given as an IV infusion at an assigned dose on Day 1 of each 21-day cycle along with either capecitabine or S-1, orally, twice daily on Days 1 to 14 of each cycle until unacceptable toxicity or symptomatic deterioration attributed to PD.
  Interventions: Drug: RO7496353; Drug: Capecitabine; Drug: S-1; Drug: Nivolumab; Drug: Oxaliplatin
- Cohort C: PDAC (Experimental): Participants with PDAC will receive RO7496353, and atezolizumab, given as an IV infusion at an assigned dose on Days 1 and 15 of each 28-day cycle along with nab-paclitaxel, and gemcitabine, also given as an IV infusion on Days 1, 8, 15 of each 28-day cycle until unacceptable toxicity or symptomatic deterioration attributed to PD.
  Interventions: Drug: RO7496353; Drug: Atezolizumab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Substudy: UC (Experimental): Participants with UC will receive RO7496353, and atezolizumab, given as an IV infusion at an assigned dose on Day 1 of each 21-day cycle until unacceptable toxicity or symptomatic deterioration attributed to PD.
  Interventions: Drug: RO7496353; Drug: Atezolizumab

INTERVENTIONS:
Drug: RO7496353 — RO7496353 will be administered as per the schedules specified in the respective arms.
  Other Names: SOF 10
Drug: Atezolizumab — Atezolizumab will be administered as per the schedules specified in the respective arms.
  Other Names: RO5541267; Tecentriq
  Arms: Cohort A: NSCLC; Cohort C: PDAC; Substudy: UC
Drug: Capecitabine — Capecitabine will be administered as per the schedule specified in the respective arm.
  Arms: Cohort B: GC
Drug: S-1 — S-1 will be administered as per the schedule specified in the respective arm.
  Other Names: Tegafur/Gimeracil/Oteracil potassium
  Arms: Cohort B: GC
Drug: Nivolumab — Nivolumab will be administered as per the schedule specified in the respective arm.
  Arms: Cohort B: GC
Drug: Oxaliplatin — Oxaliplatin will be administered as per the schedule specified in the respective arm.
  Arms: Cohort B: GC
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered as per the schedule specified in the respective arm.
  Arms: Cohort C: PDAC
Drug: Gemcitabine — Gemcitabine will be administered as per the schedule specified in the respective arm.
  Arms: Cohort C: PDAC

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of RO7496353 in combination with a checkpoint inhibitor (CPI) with or without standard-of-care (SOC) chemotherapy in participants with locally advanced or metastatic solid tumors such as non-small cell lung cancer (NSCLC), gastric cancer (GC) and pancreatic ductal adenocarcinoma (PDAC).

The substudy will evaluate the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary anti-tumor activity of RO7496353 in combination with atezolizumab in patients with locally advanced or metastatic urothelial carcinoma (UC).

The parent and substudy will be conducted in 2 stages: an initial safety run-in stage and an expansion stage.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months
* Adequate hematologic and end-organ function
* Histologically confirmed locally advanced, recurrent, or metastatic incurable solid tumor malignancy
* Measurable disease according to RECIST v1.1 on computed tomography (CT) or magnetic resonance imaging (MRI) images within 28 days prior to enrollment
* Availability of representative tumor specimens in formalin-fixed, paraffin-embedded (FFPE) blocks or at least 15 unstained slides

Exclusion Criteria:

* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, and/or radiotherapy, within 3 weeks prior to initiation of study treatment
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Positive test for human immunodeficiency virus (HIV) infection
* Positive hepatitis B surface antigen (HbsAg) test, and/or positive total hepatitis B core antibody (HbcAb) test at screening
* Positive hepatitis C virus (HCV) antibody test at screening
* Known allergy or hypersensitivity to any component of the RO7496353 formulation or any of the study drugs or their excipients

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to approximately 33 months
  AEs will be reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0).

SECONDARY OUTCOMES:
Plasma Concentration of RO7496353 | Up to approximately 33 months
Percentage of Participants With Anti-drug Antibody (ADA) to RO7496353 | Up to approximately 33 months
Confirmed Objective Response Rate (ORR) as Determined by the Investigator per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Up to approximately 33 months
Duration of Response (DOR) as Determined by the Investigator per RECIST v1.1 | Up to approximately 33 months
Progression-free Survival (PFS) as Determined by the Investigator per RECIST v1.1 | Up to approximately 33 months

OTHER OUTCOMES:
Cohort A and C: Serum Concentration of Atezolizumab | Up to approximately 33 months
Cohort A and C: Percentage of Participants With ADAs to Atezolizumab | Up to approximately 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- United States (3):
  - UCLA University of California Los Angeles, Los Angeles, California
  - Yale School of Medicine, New Haven, Connecticut
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Australia (2):
  - St Vincent'S Hospital, Darlinghurst, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
- Brazil (2):
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Hospital de Câncer de Barretos, Barretos, São Paulo
- Italy (3):
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan, Lombardy
  - Centro Ricerche Cliniche Di Verona, Verona, Veneto
- Japan (5):
  - National Cancer Center Hospital East, Chiba
  - Kanagawa Cancer Center, Kanagawa
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Tokyo
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Severance Hospital Yonsei University Health System - Clinical Trials Center Pharmacy, Seoul
- Spain (4):
  - NEXT Oncology-Hospital Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Clinica Universidad de Navarra-Madrid, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Turkey (Türkiye) (2):
  - Ankara City Hospital, Ankara
  - Dokuz Eylul Universitesi Tip Fakultesi, Lzmir

IPD SHARING:
Plan to Share IPD: No